CLINICAL TRIAL: NCT02800876
Title: Evaluation of Aortic Aneurysms With Focus on Wall Stress and Wall Rupture Risk by Computational Finite Element Analysis With Dedicated Software
Brief Title: Evaluation of Aortic Aneurysms With Focus on Wall Stress and Wall Rupture Risk
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Responsible Party: Principal Investigator, Thi Dan Linh Nguyen-Kim, Dr. med., University of Zurich
Other Study IDs: KEK-ZH-Nr. 2015-0156
Record Dates: First submitted 2016-06-08; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- asymptomatic not ruptured aneurysm: Patients with asymptomatic not ruptured aortic aneurysms greater than 3 cm who received a clinical indicated CT
  Interventions: Other: CT-acquisition
- symptomatic not ruptured aneurysm: Patients with symptomatic aortic aneurysms greater than 3 cm who received a clinical indicated CT
  Interventions: Other: CT-acquisition
- symptomatic ruptured aneurysm: Patients with symptomatic ruptured aortic aneurysms greater than 3 cm who received a clinical indicated CT
  Interventions: Other: CT-acquisition
- patients with small aneurysms: Patients with small aortic aneurysms approximately 5.5 cm, ruptured and not ruptured, who received a clinical indicated CT
  Interventions: Other: CT-acquisition

INTERVENTIONS:
Other: CT-acquisition

SUMMARY:
Retrospective study to evaluate the impact of computational wall stress analysis based on computed tomography (CT) of ruptured and not-ruptured aortic aneurysms as an additional predictor for rupture with dedicated software.

DETAILED DESCRIPTION:
In patients with known aortic aneurysm who received clinically indicated CT during a time period from 01/2004-12/2013 the CT data was evaluated with dedicated software, A4clinics, VASCOPS GmbH, Graz, Austria. The following parameters will be evaluated: exterior and luminal diameter, intraluminal thrombus (ILT) thickness, vessel-, luminal- and intraluminal thrombus volume, peak wall stress (PWS), peak wall rupture risk (PWRR), von Mises-stress and rupture risk-index in the ILT.

ELIGIBILITY:
Inclusion Criteria:

Clinical indicated CT data from patients with known aortic aneurysms.

Clinical indication was:

* Follow up CT examination by known aortic aneurysm
* Patient with known aortic aneurysm with new acute clinical symptoms
* Patients with clinical suspicion of aortic aneurysm

Exclusion Criteria:

* known exclusion criteria for CT examination as known allergy to iodine or contrast media
* known pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with known aortic aneurysms, who underwent clinical indicated CT during a time period from 01/2004-12/2013
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
To calculated the rupture risk equivalent diameter (RRED) of the aortic aneurysm and rupture risk-index in the intraluminal thrombus within the aortic aneurysm. | CT Data from 01/2004-12/2013
  By using the finite analysis from the CT data the peak wall stress (PWS), the peak wall rupture (PWRR) and the mises stress within the aortic aneurysm depending on the diameter and volume of the aortic aneurysm and of the intraluminal thrombus will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland